CLINICAL TRIAL: NCT02491502
Title: Treatment of Benign Thyroid Nodules With FastScan High Intensity Focused Ultrasound (HIFU)
Brief Title: Treatment of Benign Thyroid Nodules With FastScan HIFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU/BG/TN/FS/2015
Record Dates: First submitted 2015-06-24; First posted 2015-07-08 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Benign Thyroid Nodules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Echopulse (Experimental): Echopulse HIFU
  Interventions: Device: Echopulse

INTERVENTIONS:
Device: Echopulse — HIFU Under ultrasound guidance
  Other Names: Echopulse HIFU

SUMMARY:
This study evaluates the efficacy of the HIFU for the treatment of benign thyroid nodules with the FastScan version using assessment of patient experience and adverse event reporting.

DETAILED DESCRIPTION:
Echopulse is specially designed, manufactured and CE marked for treating benign thyroid nodules. HIFU is a completely alternative to surgery which utilizes high-energy ultrasound to deliver a large amount of sound energy to a focal point to rapidly induce tissue heating to 85-90°C.This initiates tissue coagulation followed by tissue necrosis ablating the targeted area.

In a previous european feasibility study performed at 1 site (Bulgaria), 20 benign thyroid nodules were treated. The HIFU treatment was well tolerated and showed efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient 18 years or older.
* Patient presenting with at least one thyroid nodule with no signs of malignancy:

  1. Non suspect clinically and at ultrasonography imaging
  2. Benign cytological diagnosis at FNAB (fine-needle aspiration biopsy) from the last 6 months
  3. Normal serum calcitonin
  4. No history of neck irradiation
* Normal TSH (thyroid-stimulating hormone)
* Targeted nodule accessible and eligible to HIFU
* Absence of abnormal vocal cord mobility at laryngoscopy
* Nodule diameter ≥ 10mm measured by ultrasound
* Composition of the targeted nodule(s) : predominantly solid
* Patient has signed a written informed consent.

Exclusion Criteria:

* Head and/or neck disease that prevents hyperextension of neck
* Known history of thyroid cancer or other neoplasias in the neck region
* History of neck irradiation
* Macrocalcification inducing a shadow in the thyroid significant enough to preclude the HIFU treatment
* Posterior position of the nodule if the thickness of the nodule is <15mm
* Pregnant or lactating woman
* Any contraindication to the assigned analgesia/anaesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-06; Primary Completion 2020-04 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 1 day post treatment
Number of participants with adverse events | 3 days post treatment
Number of participants with adverse events | 7 days post treatment
Change in volume of the thyroid nodule compared to Baseline at 6 months | 6 months post treatment
Change from Baseline Patient pain intensity score (100mm visual analog scale) at 1 day | 1 day post treatment
Change from Baseline Patient pain intensity score (100mm visual analog scale) at 3 days | 3 days post treatment
Change from Baseline Patient pain intensity score (100mm visual analog scale) at 7 days | 7 days post treatment
Patient satisfaction questionnaire | 6 months post treatment

SECONDARY OUTCOMES:
Number of patients with Absence of palpable lesion | 3 months post treatment
Number of patients with Absence of palpable lesion | 6 months post treatment
Patient Cosmetic evaluation measured by questionnaire | 6 months post treatment
Investigator rated evaluation of the device | Post treatment Day 0
Change from Baseline of gland vascularization at 3 months | 3 months post treatment
Change from Baseline of gland vascularization at 6 months | 6 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roussanka Kovatcheva, Prof., Principal Investigator — roussanka_kov@yahoo.com
Locations (1):
- University Hospital of Endocrinology USBALE, Sofia, Bulgaria